CLINICAL TRIAL: NCT02009995
Title: The Diabetes Aerobic and Resistance Bands Exercise (DARE-Bands) Trial
Acronym: DARE-Bands
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Ron Sigal, Professor of Medicine, Cardiac Sciences, Kinesiology and Community Health Sciences, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1026315
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus; Type 2 Diabetes Mellitus; Resistance Training; Resistance Exercise; Resistance Band; Thera-band; elastic band; exercise band
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Training (AT) only (Active Comparator): All subjects will participate in a 10-week ramp-in period with the goal of achieving 150 minutes of moderate-to-vigorous physical activity per week. Walking and jogging will be the primary modes of achieving the prescribed aerobic activity as these are the modes of aerobic exercise that are most accurately recorded by an accelerometer. Subjects will use the Rate of Perceived Exertion (RPE) to guide aerobic exercise intensity. Aerobic activity will be objectively monitored by the Technogym MyWellness Key (MWK) accelerometer, which is a lightweight device worn on the waistband.
  Interventions: Behavioral: Aerobic Training (AT)
- AT plus Primarily Home-Based Resistance Band Training (Experimental): Both of the bands + AT groups will engage in RBT 3 times per week, progressing to 3 sets of 8-12 repetitions of 12 exercises. The exercises will be: chair squat, sitting chest press, seated rear fly, seated row, overhead press, lateral raise, biceps curl, triceps extension, leg extension, hamstring curl, gluteal extension, and abdominals. The resistance band exercise sessions will be between 25-60 minutes.
  Participants in this group will attend supervised group sessions weekly in weeks 1-4, every 2 weeks in weeks 5-8, and every 4 weeks thereafter to ensure proper form and appropriate progression. Participants in this group will be responsible to complete all remaining sessions (a total of 3 per week, including supervised sessions) at home on their own time.
  Interventions: Behavioral: Aerobic Training (AT); Behavioral: AT plus Primarily Home-Based Resistance Band Training

INTERVENTIONS:
Behavioral: Aerobic Training (AT) — All subjects will participate in a 10-week ramp-in period with the goal of achieving 150 minutes of moderate-to-vigorous physical activity per week. Walking and jogging will be the primary modes of achieving the prescribed aerobic activity as these are the modes of aerobic exercise that are most accurately recorded by an accelerometer. Subjects will use the Rate of Perceived Exertion (RPE) to guide aerobic exercise intensity. Aerobic activity will be objectively monitored by the Technogym MyWellness Key (MWK) accelerometer, which is a lightweight device worn on the waistband.
Behavioral: AT plus Primarily Home-Based Resistance Band Training — The bands + AT group will engage in RBT 3 times per week, progressing to 3 sets of 10-15 repetitions of 12 exercises. The exercises will be: chair squat, sitting chest press, seated rear fly, seated row, overhead press, lateral raise, biceps curl, triceps extension, leg extension, hamstring curl, gluteal extension, and abdominals. The resistance band exercise sessions will be between 25-60 minutes.
  Participants in this group will attend supervised group sessions weekly in weeks 1-4, every 2 weeks in weeks 5-8, and every 4 weeks thereafter to ensure proper form and appropriate progression. Participants in this group will be responsible to complete all remaining sessions (a total of 3 per week, including supervised sessions) at home on their own time.
  Arms: AT plus Primarily Home-Based Resistance Band Training

SUMMARY:
BACKGROUND Resistance exercise training with free weights or weight machines clearly improves glucose (sugar) control in type 2 diabetes (T2D). However, many patients with T2D would prefer not to attend an exercise facility, for reasons of cost and/or convenience. Coinvestigator Jonathon Fowles has developed and pilot-tested a home-based exercise program for people with T2D using resistance bands. However, the effects of resistance-bands training (on glucose control in T2D have not been evaluated in a high-quality randomized trial.

SPECIFIC AIMS To determine the effects of six months of progressive home-based resistance bands training (RBT) versus no RBT in people with T2D on blood glucose control (HbA1c, primary outcome), waist circumference, heart disease risk factors, and quality of life.

METHODS A total of 100 T2D participants will be randomized to 2 arms: home-based RBT (RBT-H) or aerobic training only (ATO). Both groups will accumulate 150 minutes per week of aerobic exercise such as walking. The resistance exercise workout includes 12 exercises, targeting all major muscle groups. RBT-H subjects will complete most exercise at home with periodic supervision.

SIGNIFICANCE The global burden of type 2 diabetes is increasing, and complications of the illness occur primarily in those whose glucose control is fair or poor. If exercise training with resistance bands improves glucose control, it could be beneficial to the large numbers of patients who cannot travel to a gym or cannot afford gym membership. If resistance exercise is then adopted by more patients, it is likely that the morbidity associated with type 2 diabetes will be decreased. This is particularly true if such training also improves quality of life, and more people are thus inclined to continue exercising in the long term.

DETAILED DESCRIPTION:
BACKGROUND Resistance exercise training with free weights or weight machines clearly improves glycemic control in type 2 diabetes (T2D). However, many patients with T2D would prefer not to, or are not able to attend an exercise facility,for reasons of cost, comfort or convenience. Coinvestigator Dr. Jonathon Fowles developed a home-based exercise program for people with T2D using resistance bands. Before-after studies using this intervention have found improvements in glycemic control, strength, and blood pressure. However, the effects of resistance-bands training (RBT) on glycemic control in T2D have not been evaluated in a high-quality randomized trial.

RESEARCH QUESTIONS To determine the effects of six months of progressive home-based RBT plus aerobic exercise, versus home-based aerobic exercise alone, in previously-sedentary people with T2D.

METHODS After a 2-week run-in period to assess adherence, 100 T2D subjects not currently engaging in regular exercise will be randomized in equal numbers to 2 arms: primarily home-based RBT (RBT-H) or aerobic only control (ATO) . Both groups will complete aerobic training: accumulation of 150 minutes per week of walking or jogging, measured by accelerometers. The RBT workout will include 12 distinctive exercises, targeting all major muscle groups. Subjects will be trained in groups led by a Kinesiologist (exercise specialist) twice per week for two weeks during run-in. After randomization, the RBT-H group will perform RBT three times per week. RBT-H participants will perform RBT three times per week primarily at home, with supervised group sessions weekly in weeks 1-4, every 2 weeks in weeks 5-8, and every 4 weeks thereafter to ensure proper form and appropriate progression. Adherence to RBT will be verified through direct supervision of group sessions, and completion of detailed exercise logs for home-based and group sessions. Participants will photograph the log after each session and email the photo to a designated email address. Study outcomes will be assessed at baseline, 12 and 24 weeks post-randomization. Dietary advice will be standardized through repeated sessions with a dietician, and doses of medications altering glucose, lipids and BP will be held constant unless change is medically urgent. Primary analyses will be intention-to-treat, using repeated measures mixed modeling. Per-protocol analyses will be done including only subjects who completed >70% of prescribed exercise sessions and all end-of-study outcome measures.

SIGNIFICANCE The global burden of type 2 diabetes is increasing, and complications of the illness occur primarily in those whose glycemic control is fair or poor. If home-based exercise training with resistance bands improves glycemic control and other vascular risk factors, it could be beneficial to the large numbers of patients who prefer not to have to travel to a gym or cannot afford gym membership. If resistance exercise is then adopted by more patients, it is likely that the morbidity associated with type 2 diabetes will be decreased. This is particularly true if such training also improves quality of life, and more people are thus inclined to continue exercising in the long term.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged >35 years with T2D as defined by the CDA Expert Committee.
2. A1C values within range of 6.6%-9.9%.
3. Willingness to follow study procedures (e.g. wear the accelerometer for exercise sessions and download them at least weekly, complete exercise logs, attend supervised group-based resistance band sessions, perform resistance bands exercise at home).

Exclusion Criteria:

1. Participation in a regular program of physical conditioning or aerobic sports/activities for >150 minutes per week during the 6 months prior to enrolment.
2. Participation in any resistance exercise training during the previous 6 months.
3. Requirement for insulin therapy currently or in the previous 3 months.
4. Uncontrolled hyperglycemia (A1C > 10%), as it would be a clear indication for cointervention.
5. Uncontrolled hypertension: systolic BP >160 mmHg or diastolic BP >100 mmHg, both measured in sitting position. If too-high A1C or BP is the only reason for exclusion, subjects will be asked to see their physicians regarding the hyperglycemia or BP, and invited to re-apply for the study several months later if the problem is under better control.
6. Hypo-glycemia unawareness, or severe hypoglycemia requiring assistance from another person within the previous 3 months.
7. Restrictions in physical activity due to disease: unstable cardiac or pulmonary disease, severe aortic stenosis, Marfan's syndrome (risk of aortic dissection from resistance training), intermittent claudication sufficient to interfere with aerobic exercise progression, severe peripheral neuropathy or active proliferative retinopathy, disabling stroke, severe arthritis, musculoskeletal injuries compromising safety of the prescribed exercises, inability to walk 10 minutes.
8. Other illness, judged by the patient or study physician to make participation in this study inadvisable.
9. Inability to understand or comply with instructions.
10. Pregnancy at the start of the study, or intention to become pregnant in the next 6 months.
11. Plans to move to a different city within the next 12 months.
12. Inability to communicate in English or French.
13. Unwillingness to sign informed consent.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Testing of Strength | Baseline, 12 weeks, 24 weeks
  The maximum weight that can be lifted 8 times while maintaining proper form (8RM) will be determined for chest press (upper body) and leg press (lower body).

SECONDARY OUTCOMES:
Blood Pressure | Baseline, 12 weeks, 24 weeks
  Three measures of systolic and diastolic blood pressure (BP) will be taken at 2-minute intervals using a BP-Tru automated BP monitor (BP-Tru, Coquitlam, BC), with the subject sitting with back supported; the mean of the lower two measures will be taken as the true BP.
Smoking | baseline
  will be assessed by self-report (number of cigarettes/day). The smoking rate is expected to be low and we do not expect intergroup differences. We will gather this information because smoking, an important predictor of diabetic complications including CVD, is used in the UKPDS Outcomes Model.
Traditional lipids | Baseline, 12 weeks, 24 weeks
  Total cholesterol, HDL-Cholesterol and triglycerides will be measured by enzymatic colorimetric assays, and LDL-C calculated using the Friedewald equations. Total cholesterol/HDL-cholesterol ratio will be calculated.
Apolipoproteins | Baseline, 12 weeks, 24 weeks
  Apolipoprotein B (ApoB), Apolipoprotein A-1 (ApoA1), ApoB/ApoA1 ratio.
HSCRP | Baseline, 12 weeks, 24 weeks
  Addition of HSCRP (High-sensitivity C-reactive Protein) levels to cardiac risk prediction equations can provide incremental risk discrimination beyond that provided by age, sex, smoking, BP, and diabetes.
Moderate-vigourous aerobic exercise | every week from baseline to 24 weeks
  Weekly time spent in moderate-to-vigourous intensity physical activity (i.e. greater than 3 METs) as measured by the MyWellness Key accelerometer will be collected via the web-based interface.
The UKPDS Outcomes Model | Baseline, 12 weeks, 24 weeks
  is a computer simulation model for forecasting the occurrence of seven diabetes-related complications.
Satisfaction with the exercise program | 12 and 24 weeks
  Structured interview.
Continued participation in exercise after end of intervention | 3, 6, 9, 12, 15, 18, 21, 24 months after completion of the intervention
  telephone interviews every 3 months for 2 years after the end of the intervention period.
Medication Changes | Baseline, 12 weeks, 24 weeks
  Medication and doses will be assessed. Changes (start/increased dose; stop/decreased dose) in medications altering glucose, lipids or blood pressure will be considered secondary outcomes.
Adverse Events | Baseline, 12 weeks, 24 weeks
  Participants will be questioned regularly at each clinic visit regarding adverse events, which will be tracked systematically using standard forms.
Hemoglobin A1c (A1C) | Baseline, 12 weeks, 24 weeks
  A1C reflects average blood glucose over the previous 2-3 months and is expressed as a percent (normal A1C 4-6%, target A1C in diabetes <7%). A 1% absolute decrement in A1C (e.g. from 8.0% to 7.0%) is associated with a 37% lower risk of microvascular complications of diabetes. In epidemiological analyses, lower A1C was also associated with lower risk of CVD. There has never been a negative impact of A1C-lowering in exercise trials.
Weight | Baseline, 12 weeks, 24 weeks
  Taken in light clothing without shoes.
Waist circumference | Baseline, 12 weeks, 24 weeks
  Measured midway between the lowest rib and the top of the iliac crest.
Hip circumference | Baseline, 12 weeks, 24 weeks
  Measured around the widest portion of the buttocks.
SF-36 questionnaire | Baseline, 12 weeks, 24 weeks
  Used to assess health related quality of life.
Diabetes Distress Scale Questionnaire | Baseline, 12 weeks, 24 weeks
  Assesses emotional distress and functioning specific to living with diabetes.
EuroQOL EQ-5D questionnaire | Baseline, 12 weeks, 24 weeks
  Assesses five core domains of quality of life (mobility, self-care, ability to conduct usual activities, pain and discomfort, and anxiety and depression).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Sigal, MPH, MD, Principal Investigator — University of Calgary, Faculty of Medicine
Locations (1):
- Richmond Road Diagnostic and Treatment Centre, Calgary, Alberta, Canada